CLINICAL TRIAL: NCT03772171
Title: Evaluation of the Use of an Analog Scale to Estimate Dietary Intakes, EPA, for Hemodialysis Patients
Brief Title: Estimate for Dietary Intakes and Hemodialysis Patients
Acronym: EDDEN
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 17-250
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Nutrition Disorders; Dialysis; Chronic Renal Failure; Dietetician
MeSH Terms: conditions — Nutrition Disorders; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this clinical research is to evaluate the relevance of using the EPA slide to estimate dietary intakes in dialysis patients. The obtained results will be compared with the reference technique validated by the HAS: food intake over 3 days.

The aim is also to improve the global management of dialysis patients and improve their quality of life. The aim is to evaluate a quick and easy-to-use tool whose use has been demonstrated in hospitals but for which no study has been carried out in an ambulatory hospitalization context.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be able to understand and voluntarily sign an informed consent form
* Patient with chronic end stage renal failure treated with hemodialysis.
* Patient with age >= 18 years

Exclusion Criteria:

* Patient treated by peritoneal dialysis
* Patient with age < 18 years
* Patient with intellectual limitations that may limit the comprehension of questionnaires
* Patient with communication disorders or verbal comprehension
* Patient not French speaking
* Patient with enteral nutrition
* Patient having been hospitalized for less than 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic end stage renal failure treated by hemodialysis in hemodialysis center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of the validity of the EPA to estimate, on an outpatient basis, dietary intakes in dialysis patients | 10 days
  The Gold Standard will calculate the energy intake of the patient from the food intake over 3 days, as a percentage of its energy needs, calculated according to the weight of the patient (actual weight if weight <30kg.m² and weight adjusted if weight ≥ 30kg.m²).

CONTACTS AND LOCATIONS:
Locations (1):
- Néphrology Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided